CLINICAL TRIAL: NCT01479582
Title: A Multicenter Access and Distribution Protocol for Unlicensed Cryopreserved Cord Blood Units (CBUs) for Transplantation in Pediatric and Adult Patients With Hematologic Malignancies and Other Indications
Brief Title: Providing Access to Cord Blood Units for Transplants
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120027; 12-C-0027
Record Dates: First submitted 2011-11-22; First posted 2011-11-24 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2012-11-26

CONDITIONS: Chronic Myelogous Leukemia/Other Leukemia; Acute Leukemias; MDS/MPS; Multiple Myeloma; Non-Hodgkin Lymphoma
Keywords: Adult and Pediatric; Unlicensed Cord Blood Unit IND; NMDP; Transplant; Hematologic Malignancies; Leukemia; Multiple Myeloma; Non-Hodgkin Lymphoma; CML; Chronic Myelogenous Leukemia; Myelodyplastic Syndrome; MDS; Thalassemia; Lysosomal Storage Diseases
MeSH Terms: conditions — Multiple Myeloma; Lymphoma, Non-Hodgkin; Hematologic Neoplasms; Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Thalassemia; Lysosomal Storage Diseases

INTERVENTIONS:
Drug: Access to unlicensed cord blood units

SUMMARY:
Background:

- Cord blood banks have been set up to collect and store umbilical cord blood for transplants. These transplants are used to treat different types of cancer. In October 2011, the Food and Drug Administration (FDA) began considering cord blood as a biological drug. Most of the cord blood units currently available in cord blood banks in the United States and other countries were collected before the FDA set these new standards. The units meet standards set by the National Marrow Donor Program (NMDP), but they were not collected, tested, or stored exactly according to FDA standards. As a result, the new guidelines state that they may only be used for transplant if the transplant is done as part of a study. Researchers have set up a study to provide these cord blood units to recipients and to study the effects of their use.

Objectives:

* To provide access to cord blood units for recipients whose best choice for a unit meets NMDP but not FDA standards.
* To study the effects of these cord blood transplants.

Eligibility:

- Individuals who need to have a cord blood transplant to treat certain types of cancer.

Design:

* Participants will be screened with a physical exam, medical history. They will also have blood tests and imaging studies.
* Participants will have the cord blood transplant and allow their medical data to be collected by the study researchers.

DETAILED DESCRIPTION:
Study Design:

This study is an access and distribution protocol for unlicensed cryopreserved cord blood units (CBUs) in pediatric and adult patients with hematologic malignancies and other indications.

Primary Objective:

The primary aim of this study is to examine the incidence of neutrophil recovery of (Bullet)500/mm3

after cord blood transplantation in a multi-institution setting using CBUs that are not Food and

Drug Administration (FDA) licensed.

Secondary Objectives:

In patients receiving a non-licensed CBU:

* Assess incidence of graft rejection
* Assess incidence of transmission of infection
* Assess incidence of serious infusion reaction
* Determine 1 year survival after cord blood transplantation
* Assess cumulative incidence of acute graft vs. host disease (GVHD) grades II to IV and

grades III to IV

* Assess cumulative incidence of chronic GVHD
* Determine platelet engraftment of >20,000 mcL and >50,000 mcL
* Determine CBU-derived engraftment

Eligibility Criteria:

Inclusion Criteria

* Patients with FDA-specified indications (see Appendix B for further details):
* Hematological malignancies
* Certain lysosomal storage and peroxisomal enzyme deficiency disorders
* Hurler syndrome (MPS I)
* Krabbe Disease (Globoid Leukodystrophy)
* X-linked Adrenoleukodystrophy
* Primary immunodeficiency diseases
* Bone marrow failure
* Beta-thalassemia
* Signed informed consent (and signed assent, if applicable)
* Pediatric and adult patients of any age

Exclusion Criteria

* Patients who are receiving only licensed CBUs
* Cord blood transplant recipients at international transplant centers

Treatment Description:

Treatment, including pre-transplant conditioning and GVHD prophylaxis, will occur per each

transplant center s specifications.

Accrual Objective:

In this access and distribution protocol, U.S. patients undergoing transplant using unlicensed

CBUs will be enrolled and there is no accrual maximum.

Accrual Period:

The accrual period is open ended.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients with FDA-specified indications:

* Hematological malignancies
* Certain lysosomal storage and peroxisomal enzyme deficiency disorders
* Hurler syndrome (MPS I)
* Krabbe Disease (Globoid Leukodystrophy)
* X-linked Adrenoleukodystrophy
* Primary immunodeficiency diseases
* Bone marrow failure
* Beta-thalassemia
* Signed informed consent (and signed assent, if applicable)
* Pediatric and adult patients of any age

EXCLUSION CRITERIA:

* Patients who are receiving only licensed CBUs
* Cord blood transplant recipients at international transplant centers

Max Age: 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2011-10-27; Primary Completion 2012-11-26 (Actual); Study Completion 2012-11-26 (Actual)

PRIMARY OUTCOMES:
The primary aim of this study is to examine the incidence of neutrophil recovery of greater than or equal to 500/mm3 after cord blood transplantation in a multi-institution setting using CBUs that are not Food and Drug Administration (FDA) licen...

SECONDARY OUTCOMES:
Assess incidence of graft rejection.
Assess incidence of transmission of infection.
Assess incidence of serious infusion reaction.
Determine 1 year survival after cord blood transplantation.
Assess cumulative incidence of aGVHD vs cGVHD.

CONTACTS AND LOCATIONS:
Overall Officials: Ronald E Gress, M.D., Principal Investigator — National Cancer Institute (NCI)

REFERENCES:
- [Background] Laughlin MJ, Barker J, Bambach B, Koc ON, Rizzieri DA, Wagner JE, Gerson SL, Lazarus HM, Cairo M, Stevens CE, Rubinstein P, Kurtzberg J. Hematopoietic engraftment and survival in adult recipients of umbilical-cord blood from unrelated donors. N Engl J Med. 2001 Jun 14;344(24):1815-22. doi: 10.1056/NEJM200106143442402. PMID 11407342
- [Background] Kurtzberg J, Laughlin M, Graham ML, Smith C, Olson JF, Halperin EC, Ciocci G, Carrier C, Stevens CE, Rubinstein P. Placental blood as a source of hematopoietic stem cells for transplantation into unrelated recipients. N Engl J Med. 1996 Jul 18;335(3):157-66. doi: 10.1056/NEJM199607183350303. PMID 8657213
- [Background] Rocha V, Labopin M, Sanz G, Arcese W, Schwerdtfeger R, Bosi A, Jacobsen N, Ruutu T, de Lima M, Finke J, Frassoni F, Gluckman E; Acute Leukemia Working Party of European Blood and Marrow Transplant Group; Eurocord-Netcord Registry. Transplants of umbilical-cord blood or bone marrow from unrelated donors in adults with acute leukemia. N Engl J Med. 2004 Nov 25;351(22):2276-85. doi: 10.1056/NEJMoa041469. PMID 15564544